CLINICAL TRIAL: NCT05051839
Title: Randomized Clinical Trial to Validate Use of Implants and Abutments With Biologically Oriented Preparation Technique (I.B.O.P.T.)
Brief Title: Validation Use of Implants and Abutments With Biologically Oriented Preparation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14/532
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Dental Implant-Abutment Design

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiographic bone level (Experimental)
  Interventions: Procedure: Implant surgery and restoration
- Peri implant soft tissue volume (Experimental)
  Interventions: Procedure: Implant surgery and restoration

INTERVENTIONS:
Procedure: Implant surgery and restoration — Implants with two different transmucosal neck configuration are placed.

SUMMARY:
This randomized clinical trial aims to validate and to establish indications for using implants with biological oriented preparation technique (I.B.O.P.T.) for implant supported prosthetic treatment as an option looking for better stability and control of associated soft and hard tissues compared with conventional implants and conventional abutments with finishing lines preparation technique.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old.
* Need for implant-supported fixed prosthesis in the posterior area of the upper or lower jaw (up to 2 implants and three units bridge);
* Adequate bone quality and quantity at the implant site to allow the insertion of Sweden and Martina Premium or Prama (Due Carrare, Padova, Italy), of diameters 3.8, 4.25 or 5 mm and lengths between 10 and 13 mm.
* Healthy ASA type I and II patients.
* Full-mouth plaque index <20.

Exclusion Criteria:

* Smokers ≥10 cigarettes/day.
* Presence of implant-supported restorations adjacent to the study site.
* Active periodontitis defined as the presence of pockets with probing depth (PD) ≥5 mm and bleeding on probing (BoP).
* Systemic medication that contraindicates surgery (bisphosphonates or steroid therapy).
* Uncontrolled diabetes.
* Severe bruxism.
* Pregnancy.
* Previous history of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Marginal bone level | Baseline to 12-months follow-up
  Changes in interproximal marginal bone level with standardization of the radiograph
Soft tissue volumetric analysis | Baseline to 12-motnhs follow-up
  Soft tissue volumetric analysis with digital impressiones taken at baseline and at 12-month follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Unviersidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No